CLINICAL TRIAL: NCT01435421
Title: Breath Test for Patients With Acute Liver Disease for Early Detection of the Need for Transplant or Recovery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: ALF-BID-1108-HMO-CTIL
Record Dates: First submitted 2011-09-15; First posted 2011-09-16 (Estimated); Last update posted 2011-09-16 (Estimated); Status verified 2011-09

CONDITIONS: Acute Liver Failure
MeSH Terms: conditions — Liver Failure, Acute

SUMMARY:
Acute liver failure (ALF) results from an abrupt loss of hepatic metabolic and synthetic function and leads to encephalopathy and potentially multi-organ dysfunction. Aetiologies include autoimmune and metabolic diseases, infectious agents and hepatotoxins. Worldwide, infectious hepatitis (A, B and E) is the most common cause. In Western Europe and the USA, ALF is most frequently caused by paracetamol intoxication.

The MBT can produce immediate results to aid in decision making in patients with acute liver disease. Such a test may affect decision-making regarding transplantation in this setting, facilitate appropriate discharge from critical care to other hospital units and to home, provide point of care assessment of therapeutic interventions.

The BreathID can potentially help in determining:

* Parameter to include patients in transplant list (the UNOS 1A group)
* Identification that patient deteriorates and needs extended hospitalization/referral to ICU/change in management
* An addition to the MELD and or other scores to estimate risk in other acute patients
* Additional information to that of other commonly utilized prognostic scoring systems

The primary end-point of the study is to develop a model to predict deterioration of the liver disease, which incorporates measurements from the MBT along with other potential variables. The data collected will be used to develop a prediction model using data-mining methodology (linear and non-linear regression models, binary trees, neural networks, etc…). The predictive models may include measurements from the MBT, blood test results, as single measurements or as trend over time. The model that will be developed, will attempt to predict the disease deterioration vs. recovery accurately, at an earlier time point than the standard procedure. A threshold will then be determinate based on adequate sensitivity and specificity levels.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men or women (>18 years of age).
2. Acute Liver insult
3. No evidence of cirrhosis (unless clinical acute Wilsons)
4. INR > 1.5
5. Duration of illness < 24 weeks -

Exclusion Criteria:

1. Patient with any chronic liver disease
2. Patient has severe congestive heart failure
3. Patient has severe pulmonary hypertension
4. Patient has chronic renal insufficiency with severe cardiac disease
5. Patient has previous surgical bypass surgery for morbid obesity
6. Patient has extensive small bowel resection
7. Patient with established extra-hepatic auto-immune disease on long term treatment
8. Patient is a recipient of any organ transplant (within the last 3 months)- Patient with proven or suspected hepatocellular carcinoma
9. Patient is pregnant
10. Patient allergic to paracetamol (such as Tylenol or any other related medications)
11. Patients in whom oral intake is contra-indicated
12. Patient, based on the opinion of the investigator, should not be enrolled into this study
13. Patients or their nominated representative is unwilling to sign informed consent
14. Patients that are participating in other clinical trials evaluating experimental treatments or procedures, not including observatory trials -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that are hospitalaized.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-12 (Estimated)